CLINICAL TRIAL: NCT03115151
Title: A Comparison of Epidural and Intravenous Patient-Controlled Analgesia Following Lumbar Spinal Fusion Surgery: A Prospective Randomized Study
Brief Title: Epidural and Intravenous Patient-Controlled Analgesia Following Lumbar Spinal Fusion Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The surgical team has difficulty to find level 1 and 2 fusions for the study.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Enas Kandil, ASSOC PROFESSOR - Anesthesiology & Pain Mgmt, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 092016-061
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Results first posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Bupivacaine; Hydromorphone; Fentanyl; Analgesics, Opioid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Patient-Controlled Epidural Analgesia (Experimental): Bupivacaine and fentanyl infusion via Continuous Lumbar Epidural Analgesia during postoperative 72 hours
  Interventions: Drug: Bupivacaine; Drug: Fentanyl
- Intravenous patient-controlled analgesia (Sham Comparator): Postoperative intravenous patient-controlled analgesia (IV PCA) with Hydromorphone
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Bupivacaine — Bupivacaine (0.0625%) will be combined with fentanyl for postoperative epidural analgesia via a lumbar epidural catheter
  Other Names: Bupivacaine Hydrochloride
  Arms: Patient-Controlled Epidural Analgesia
Drug: Hydromorphone — Hydromorphone will be given continuous infusion for intravenous patient controlled analgesia (syringe 25 mg/50 mL).
  Other Names: DILAUDID
  Arms: Intravenous patient-controlled analgesia
Drug: Fentanyl — Fentanyl (2 mcg/ml) will be given via epidural route together with bupivacaine.
  Other Names: Opioid
  Arms: Patient-Controlled Epidural Analgesia

SUMMARY:
Postoperative analgesia following spine surgery is difficult to manage. Current treatment modalities rely heavily on opioid analgesics with all of the inherent limitations and side effects. While current best practice focuses on a 'multimodal approach' (i.e. using multiple different drugs and techniques to control pain after surgery), there is no consensus regarding which components of this multimodal therapy provide optimal analgesia. This prospective randomized study will enroll patients undergoing elective Lumbar Spinal Fusion Surgery at Zale Lipshy University Hospital. The primary objective is to determine the comparative efficacy of epidural analgesia, as compared with intravenous (IV) patient-controlled analgesia (PCA), on post-operative analgesia.

DETAILED DESCRIPTION:
Study Design: Prospective study of 58 subjects undergoing elective Lumbar Spinal Fusion (1-3 levels- posterior approach) at UTSW Zale Lipshy University Hospital with:

1. Continuous Lumbar Epidural Analgesia (Patient-Controlled Epidural Analgesia- PCEA groups)
2. Intravenous Patient-Controlled Analgesia (IV PCA)

Study Interventions - The intervention to be evaluated in this study is epidural analgesia using an infusion of 0.0625% bupivacaine plus fentanyl 2mcg/ml. The epidural infusion will be continued until it is appropriate to transition the patient to a regimen of oral pain medications. Duration of epidural catheter will be 72 hours a postoperatively.

For subjects in the IV PCA group, the intervention will include post-operative IV PCA with Hydromorphone.

Epidural catheters will be placed by the spine surgeon under direct visualization intra-operatively prior to closing the surgical incision. Intra-operative epidural catheter placement by the spine surgeon will typically be done at the upper end of the dural exposure/laminectomy.

Epidurals will be assessed for efficacy/function in the recovery room post-operatively by the APS, and then daily on the floor post-operatively (unless contacted by the floor nurse regarding specific concerns).

Visual analog pain scale (VAS) will be used to evaluate degree of pain at 3, 24, 48, and 72 hours after surgery.

Additionally, both the IV PCA and the epidural PCEA groups may be given additional "rescue" pain medications as needed in the recovery room, and these may be continued through the post-operative period on the floor.

Total study duration is approximately 50 days, which starts from operating room admission for spinal fusion surgery to the first follow-up visit after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects aged 18 years or older
* Scheduled for elective posterior lumbar spinal fusion surgery between 1 and 3 levels

Exclusion Criteria:

* Baseline cognitive deficits sufficient to make objective pain self-assessments unreliable in the estimation of the Study Investigators.
* Immunocompromised subject
* Coagulopathy
* Severe liver and renal dysfunction
* Preoperative neurological deficits
* The dura damage during surgery
* Inability to follow directions or comprehend the English language.
* Females who are pregnant as determined by positive pregnancy test on or before the day of surgery.
* Prisoners.
* Patient refusal to provide informed consent.
* Allergy to amide local anesthetics (lidocaine, bupivacaine, ropivacaine) or opioid (fentanyl) allergy if patient assigned epidural analgesia.
* Hydromorphone allergy if patient assigned IV PCA

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2023-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enas Kandil, MD, Study Chair — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University Of Texas Southwestern Medical Center, Zale University Hospital, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patient-Controlled Epidural Analgesia | Intravenous Patient-controlled Analgesia
Started | 23 | 23
Completed | 17 (Study closed because study surgeon left the Institution) | 18 (Study closed because study surgeon left the Institution)
Not Completed | 6 | 5
Not completed — Intervention discontinue due to clinical condition | 2 | 2
Not completed — Epidural catheter removal | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Intervention not received according to the protocol. | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Randomization not applied | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient-Controlled Epidural Analgesia | Intravenous Patient-controlled Analgesia | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Categorical [Count of Participants; unit: Participants] — Year Population: Analysis sample is lower than total enrollment number because all participants could not completed study.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 5 | 9 | 14
    >=65 years | 12 | 9 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] — Years
  years | 66.8 (6) | 60 (14) | 63.37 (11.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 26
  Male | 6 | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 16 | 17 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 14 | 16 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Preoperative Pain Score [Mean (Standard Deviation); unit: units on a scale (0 to 100)] — VAS pain score on the scale of 0 to 100 (0=no pain, 100= worst pain)
  units on a scale (0 to 100) | 39.47 (23.09) | 35.38 (26.40) | 37.37 (24.57)

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Pain Score (VAS)
Description: Postoperative Visual Analog Pain Score following lumbar fusion surgery. VAS on the scale 0 to 100 (0= no pain, 100= worst pain).
Time Frame: VAS score at postoperative 24 hours
Population: Spinal fusion surgeries level 1 to 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient-Controlled Epidural Analgesia | Intravenous Patient-controlled Analgesia
Number analyzed (Participants) | 17 | 18
units on a scale | 40.23 (24.69) | 54.27 (25.41)

ADVERSE EVENTS:
Time Frame: All unexpected or serious adverse events have been monitored during hospital stay and 6-week follow-up period.
Arm/Group | Patient-Controlled Epidural Analgesia | Intravenous Patient-controlled Analgesia
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 0/19 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT03115151/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-08): https://cdn.clinicaltrials.gov/large-docs/51/NCT03115151/ICF_001.pdf